CLINICAL TRIAL: NCT01733134
Title: Acute Heart Failure With High Copeptin Levels Treated With Tolvaptan Targets Increased AVP Activation for Treatment Efficacy
Brief Title: Acute Heart Failure Patients With High Copeptin Treated With Tolvaptan Targets Increased AVP Activation for Treatment (ACTIVATE)
Acronym: ACTIVATE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to quit funding before any enrollments
Sponsor: Maisel, Alan, M.D. (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry); Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTIVATE117
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2016-09

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure; emergency department; copeptin; adh antagonists
MeSH Terms: conditions — Emergencies; Diabetes Insipidus | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard therapy plus Tolvaptan (Experimental): Patient in the interventional group will receive tolvaptan in addition to standard therapy
  Interventions: Drug: Tolvaptan
- Standard therapy plus placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan 30 mg. tablet for subjects enrolled prior to first 8 hours of coming to an emergency department. Repeated daily up to 5th day.
  Other Names: Samsca
  Arms: Standard therapy plus Tolvaptan
Drug: placebo — Patient in the placebo group will receive tolvaptan in addition to standard therapy
  Arms: Standard therapy plus placebo

SUMMARY:
Patients being hospitalized for acute heart failure and already receiving standard therapy will be randomized to receive either tolvaptan or placebo, based on the level of copeptin measured in their bloodstream. Patients with high copeptin levels will be able to participate in the trial, patients with low levels will be excluded. Patients being admitted to the observation unit for acute heart failure and already receiving standard therapy will be randomized to receive either tolvaptan or placebo without consideration of the copeptin level. The hypothesis is that patients receiving tolvaptan will have better improvement of shortness of breath than those receiving placebo, within 9 hours of drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Older than or equal to 18 years of age, with diagnosis and planned treatment for Acute Heart Failure
2. Dyspnea at rest or minimal exertion per the patient
3. Evidence of extracellular volume expansion by at least one of the following: JVD, Rales, Ascites, Edema or positive Chest X-ray defined as cardiomegaly, pulmonary vascular congestion, Kerley B-lines, pulmonary edema and/or pleural effusion.
4. Elevated BNP level >200 pg/ml, or NTproBNP > 1000pg/mL
5. Able to administer study drug within 8 hours from triage time

Inpatient Hospitalized Inclusion Only:

Co-peptin level > 27 pmol/L

Exclusion Criteria:

1. Unable to provide informed consent
2. Unable to have 30 day telephone follow up
3. Not expected to survive past 6 months
4. On Renal replacement therapy or creatinine >3.5
5. History of allergy or intolerance to Tolvaptan
6. Suspected Pregnancy
7. Cardiogenic Shock
8. Participation in any interventional trial in prior 30 days.
9. Receiving or planned to receive IV Inotropic therapy
10. ACS now or in the past 30 days
11. Treatment with IV infusion vasoactive drugs in the hour prior to enrollment
12. Temperature > 100.5
13. Heart Failure due to atrial fibrillation with Rapid Ventricular Response
14. SBP < 90 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Dyspnea | 9 hours
  Dyspnea will be evaluated at 9 hours

SECONDARY OUTCOMES:
Length of stay | during hospitalizaton
  The length of hospitalization will be compared between the placebo and interventional cohorts
Rehospitalization | 30 days
  The number and length of re-hospitalizations will be compared between the placebo and interventional cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Maisel, MD, Principal Investigator